CLINICAL TRIAL: NCT03171181
Title: Unilateral Peripheral Vestibular Dysfunction: Reeducation and Spatial Orientation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Aragon Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Pilar Dominguez-Olivan, Ph D. Physical Therapist., Universidad de Zaragoza
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Universidad de Zaragoza
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Inner Ear Disease; Equilibrium; Disorder, Labyrinth; Spatial Navigation
Keywords: Spatial cognition, vestibular system, motor control
MeSH Terms: conditions — Labyrinth Diseases; Spatial Navigation

STUDY DESIGN:
Intervention Model Description: Longitudinal case-control study. Accidental sampling. Single - centre study (Hospital Universitario Miguel Servet, Zaragoza. Spain)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UPVD non compensated (Experimental): Intervention group: 30 participants with unilateral peripheral vestibular disorders. Exposed to vestibular reeducation.
  Interventions: Other: Vestibular reeducation
- control group (No Intervention): Control group, to obtain reference values.
- UPVD compensated (No Intervention): Registered spatial orientation in a group of 30 participants with compensated lesion.

INTERVENTIONS:
Other: Vestibular reeducation — Balance quality was registered with static and dynamic posturography. For spatial orientation is was registered Visual vertical and visual orientation perception. Vestibular disability was also assessed. Variables were registered at the beginning and at the end of a vestibular rehabilitation in UPVD participants. Vestibular rehabilitation consisted of 10 sessions of vestibular rehabilitation using dynamic posturography and visual reeducation. Duration of each session: 40 minutes. Twice a week.
  Arms: UPVD non compensated

SUMMARY:
Motor control includes postural control and voluntary movement. For an optimal motor control it is necessary that brain integrates vestibular, visual and somatosensorial inputs properly, in a nonlinear way. Vestibular system, as an afferent organ, encodes head position in relation to gravity and changes in its linear and angular acceleration. As vestibular central system, it plays an essential role in motor control and in orientation and spatial memory as well.

When a peripheral vestibular lesion occurs, elaboration, interpretation and processing of inputs are deficient and therefore motor control is altered to a greater or lesser degree. As process progress in time, there is a natural neuroplasticity that facilitates recovery or compensate vestibular function, although sometimes this process is incomplete and requires vestibular reeducation This study aims to assess changes in balance control, orientation and handicap perception in one case group with symptomatic unilateral peripheral vestibular dysfunction, before and after a rehabilitation programme (RV). To compare values obtained at the beginning and at the end of RV to those achieved by control group. Finally, this research aims to analyse evolution of spatial orientation quality in symptomatic and non symptomatic participants.

DETAILED DESCRIPTION:
Intervention group: 30 people with a unilateral peripheral vestibular disorder (UPVD). Process lasting more than three months and symptomatic. Aged 18-66 years old.

Control group: 30 participants without UPVD, healthy for the purpose of study. No intervention group: 30 people with a unilateral peripheral vestibular disorder without symptomatology. Both groups also aged 18-66.

Balance quality was registered with static and dynamic posturography. For spatial orientation is was registered Visual vertical and visual orientation perception. Vestibular disability was also assessed. Variables were registered at the beginning and at the end of a vestibular reeducation in UPVD participants. Vestibular reeducation consisted of 10 sessions of vestibular rehabilitation using dynamic posturography and visual reeducation. Duration of each session: 40 minutes. Twice a week.

The aim is to compare data before and after intervention with those obtained in compensated patients and control group.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed of UPVD
* Length of process superior to three months
* Normal vision or corrected by lens or glasses.

Exclusion Criteria:

* Dizziness or balance alteration due to visual problem or lesion of CNS (central nervous system).
* Balance disturbance due to a locomotor cause
* Balance perturbation next to resolve.
* Sharpening or acute phase os symptoms.
* Difficulties with understanding commands.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in Visual vertical and visual orientation degrees at baseline and before treatment. | Outcomes were measured in patients at baseline and 3 months. Control group and compensated group were registered at baseline.
  Visual vertical and visual orientation were measured with bucket test

SECONDARY OUTCOMES:
Balance quality. | Outcomes were measured in patients at baseline and 3 months. Control group was registered at baseline.
  Balance quality was obtained from static and dynamic posturography

OTHER OUTCOMES:
Dizziness handicap inventory test. | Outcomes were measured in patients at baseline and 3 months.
  Quality of life was registered with Dizziness handicap inventory test (DHI).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Bengoetxea-Arrese, PhD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Facultad de Ciencias de la Salud, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are: age, sex, side of lesion and pathology. Patients are coded, so name is only known by person who makes clinical registration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2014-2018
Access Criteria: affiliation code. The rest of information is shared.